CLINICAL TRIAL: NCT05687162
Title: Brief Internet Interventions to Support Mental Health
Brief Title: SSIs for Mental Health and Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Jacobs Foundation (Unknown)
Responsible Party: Principal Investigator, Stephen Matthew Schueller, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1253
Record Dates: First submitted 2022-11-29; First posted 2023-01-18 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Loneliness; Mental Health Issue; Distress, Emotional; Depression; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Methods; abacavir

STUDY DESIGN:
Intervention Model Description: In each study, participants will be randomly assigned to complete one of three online programs, assessing DVs at baseline and 4 and 8 weeks later.
  Note that studies 1-3 have 3 arms, and study 4 has 2 arms, so in total 11 arms are included in this project.
Who Masked: Participant, Investigator
Masking Description: Participants will not be informed which condition they were assigned to or what the other conditions involve. The investigators will not interact with participants or see which condition they are in during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- (Study 1) 3-week Loneliness Program (Active Comparator): The second and third sessions are completed in the second and third week, respectively, after beginning the study.
  Interventions: Behavioral: Overcoming Loneliness three-week intervention
- (Study 1) Single-session loneliness program (Experimental)
  Interventions: Behavioral: Overcoming Loneliness single-session intervention
- (Study 1) Single-session active control program (Active Comparator)
  Interventions: Behavioral: Single-session "Sharing Feelings" program
- (Study 2) Popular online content-based single-session intervention for distress (Experimental)
  Interventions: Behavioral: The Blu Surfer program: a popular online content-based intervention for psychological distress
- (Study 2) Researcher-created single-session intervention for distress (Active Comparator)
  Interventions: Behavioral: The Action Brings Change (ABC) Program (TEAM Lab version)
- (Study 2) Online help-seeking as usual (Active Comparator)
  Interventions: Behavioral: Online help-seeking as usual
- (Study 3) Popular online content-based single-session intervention for loneliness (Experimental)
  Interventions: Behavioral: The Lonely Blu Surfer program: a popular online content-based intervention for loneliness
- (Study 3) Researcher-created single-session intervention for loneliness (Active Comparator)
  Interventions: Behavioral: Overcoming Loneliness single-session intervention
- (Study 3) Single-session active control program (Active Comparator)
  Interventions: Behavioral: Single-session "Sharing Feelings" program
- (Study 4) 23-minute loneliness program (Active Comparator)
  Interventions: Behavioral: Overcoming Loneliness single-session intervention
- (Study 4) 8-minute loneliness program (Experimental)
  Interventions: Behavioral: Overcoming loneliness SSI 8-minute version

INTERVENTIONS:
Behavioral: Overcoming Loneliness three-week intervention — A self-guided online loneliness intervention with three 10-20 minute sessions. The intervention content draws heavily from Internet Cognitive Behavioral Therapy for Loneliness and follows the form of single-session mental health interventions.
  Arms: (Study 1) 3-week Loneliness Program
Behavioral: Overcoming Loneliness single-session intervention — The Overcoming Loneliness Three-Week Intervention condensed into a single-session intervention lasting 20-30 minutes.
  Arms: (Study 1) Single-session loneliness program; (Study 3) Researcher-created single-session intervention for loneliness; (Study 4) 23-minute loneliness program
Behavioral: Single-session "Sharing Feelings" program — A self-guided online supportive therapy intervention with a single 20-30 minute session intended to encourage users to share feelings with close others. Slightly modified from the "Sharing Feelings" intervention
  Arms: (Study 1) Single-session active control program; (Study 3) Single-session active control program
Behavioral: The Blu Surfer program: a popular online content-based intervention for psychological distress — The Blu Surfer Program is a 25-minute SSI the research team developed centered on popular online content relevant to mental health. In the SSI, the user is first asked to select the kinds of support they would like to view. Next, the user is asked to explore a library of annotated popular online content (filtered by their desired kinds of content) and to select the content they find personally valuable. Finally, the SSI provides the user an annotated list of the content they selected. Users can keep this list to draw from, build on, or share later on as they wish.
  Arms: (Study 2) Popular online content-based single-session intervention for distress
Behavioral: The Action Brings Change (ABC) Program (TEAM Lab version) — The ABC project is a 20-30-minute SSI for teens based on behavioral activation. It was found to be efficacious for reducing depression, anxiety, hopelessness, and self-hate and increasing perceived control and agency in youth (link to SSI: https://osf.io/ch2tg/, license: http://creativecommons.org/licenses/by-nc-sa/4.0/). The researchers modified the phrasing in the intervention to make it more relevant to both teens and adults, as the original was designed for only teens.
  Arms: (Study 2) Researcher-created single-session intervention for distress
Behavioral: Online help-seeking as usual — This intervention, created by the present research team, aims to emulate how one might find support on their own using the internet. In this condition, participants are asked to browse the internet for 25 minutes to find popular online content relevant to their personal struggles and create an annotated list of links to the content they find useful. The intervention is similar to a "self-study" condition, which found self-study and a video intervention equally increased mental health knowledge. The survey platform provides text entry boxes to help each participant create their guide and then provides a text version of their guide for them to keep.
  Arms: (Study 2) Online help-seeking as usual
Behavioral: The Lonely Blu Surfer program: a popular online content-based intervention for loneliness — The Lonely Blu Surfer Program is a 25-minute SSI the research team developed centered on popular online content relevant to loneliness. In the SSI, the user is first asked to select the kinds of support they would like to view. Next, the user is asked to explore a library of annotated popular online content (filtered by their desired kinds of content) and to select the content they find personally valuable. Finally, the SSI provides the user an annotated list of the content they selected. Users can keep this list to draw from, build on, or share later on as they wish.
  Arms: (Study 3) Popular online content-based single-session intervention for loneliness
Behavioral: Overcoming loneliness SSI 8-minute version — A shortened version of an online self-guided intervention based on principles of CBT for loneliness. The research team created this intervention by cutting lengthy didactic material and exercises from the 23-minute version, while maintaining its core concepts.
  Arms: (Study 4) 8-minute loneliness program

SUMMARY:
This project includes three studies that explore the effectiveness of brief internet interventions for mental health and loneliness.

Study 1: The goal of this clinical trial is to examine if a brief online single-session intervention (SSI) adapted from an evidence-based internet cognitive behavioral therapy can reduce feelings of loneliness in people aged 16 and older who struggle with loneliness. The main question it aims to answer is if a brief SSI is sufficient to meaningfully reduce loneliness compared to an active control. Researchers will test these questions by comparing change in loneliness after 8 weeks between participants randomly assigned to either 1) a 30-minute online SSI for loneliness or 2) a 3-session online intervention for loneliness or 3) an active control SSI.

Study 2: The goal of this clinical trial is to examine if an SSI for psychological distress that uses popular online content as its primary form of intervention content can reduce feelings of psychological distress in people aged 16 and older who struggle with psychological distress. The main questions it aims to answer are 1) if curated popular online content can be more effective in supporting people struggling with psychological distress than researcher-created content and 2) if curated popular online content can be more effective in supporting people struggling with psychological distress than un-curated self-selected popular online content. Researchers will test these questions by comparing change in distress after 8 weeks between participants randomly assigned to either 1) 25-minute popular online content-based SSI for distress or 2) an effective 25-minute online SSI for distress with evidence-based researcher-created content or 3) online help-seeking as usual.

Study 3: The goal of this clinical trial is to examine if an SSI for loneliness that uses popular online content as its primary form of intervention content can reduce feelings of loneliness in people aged 16 and older who struggle with loneliness. The main questions it aims to answer are 1) if curated popular online content can be more effective in supporting people struggling with loneliness than researcher-created content, 2) if curated popular online content can be more effective in supporting people struggling with psychological distress than an active control, and 3) replicating the comparison in study 1, if a brief SSI is sufficient to meaningfully reduce loneliness compared to an active control. The study will test these questions by comparing change in loneliness after 8 weeks between participants randomly assigned to either 1) a 25-minute popular online content-based SSI for loneliness or 2) a 25-minute online SSI for loneliness with evidence-based researcher-created content or 3) an active control SSI.

Study 4: This experiment compared the loneliness SSI from study 1 to a version of it that lasted about half as long. It used a two-group repeated-measures experimental design, examining between-subjects differences in loneliness between baseline and eight-week follow-up between conditions.

DETAILED DESCRIPTION:
Study 1: Severe loneliness is globally prevalent and is strongly associated with impaired mental and physical well-being, making it a significant public health issue. Evidence-based interventions for loneliness reach a small subset of people who might benefit from them, so identifying new strategies for addressing loneliness at scale should be a high priority. Online single-session interventions (SSIs) have demonstrated particular promise to offer efficient and highly-scalable support to diverse populations.

The study will test if an internet-mediated self-guided SSI can produce lasting improvements in loneliness. The investigators adapted a 9-week online loneliness intervention into a 3-week 3-session version and a single-session 30-minute SSI version. The investigators will randomly assign participants to complete the 3-week version, the SSI version, or a control SSI.

The investigators will collect self-report measures at baseline, directly after the intervention, and 4 and 8 weeks after baseline. The investigators will also measure participant engagement with the intervention using self-report and behavioral measures. The investigators will recruit teens and adults (16+) for the study via social media.

Study 2: SSIs for mental health have shown promise for delivering efficient support to diverse populations. Despite their brevity, existing SSIs still struggle to engage users.

This study will explore using a broad range of mental health-relevant popular online content (eg, psychology lectures on YouTube, Instagram posts from self-care influencers, and blog posts written by people who struggle with mood disorders) in SSIs. Although it is often not evidence-based, popular online content may be more appealing and tailored to particular audiences than the researcher-created intervention content typically used in evidence-based SSIs.

In this study, researchers will examine the effectiveness of this content for addressing psychological distress. Researchers will conduct an experiment to compare a popular online content-based SSI to one that has already demonstrated efficacy and to online help seeking as usual to identify whether such content is useful within an SSI context. Researchers will measure change in psychological distress from baseline to 4-week and 8-week follow-ups.

Study 3: In this study, researchers aim to replicate and extend studies 1 and 2 to further evaluate the potential of an SSI for loneliness and the utility of popular online content as a mental health intervention.

In this study, researchers will examine the effectiveness of popular online content for addressing loneliness. Researchers will conduct an experiment to compare a popular online content-based SSI for loneliness to another online SSI for loneliness with researcher-created content and to an active control SSI. Researchers will measure change in loneliness from baseline to 4-week and 8-week follow-ups.

Study 4: This experiment tested whether a 10-minute SSI for loneliness would be less effective than a 20-minute SSI conveying the same general information. Moreover, the research team was interested in whether users would find the 10-minute version more acceptable and engaging. The research team used a two-group repeated-measures experimental design, examining between-subjects differences in change in DVs across time between conditions.This experiment was prospectively pre-registered on the Open Science Framework (https://osf.io/8bth2)

ELIGIBILITY:
Inclusion Criteria:

* Be fluent in English
* Be 16 years old + (participants in studies 2-4 recruited on CloudResearch Connect had to be at least 18)
* Have internet access and a computer, smartphone, or tablet
* To be compensated for participation and be included in the main analysis, participants in studies 1 and 2 must meet criteria for "struggling with loneliness" (ie, a score on the 3-item loneliness screen of at least 6, and indicating that one's loneliness is causing one distress). Otherwise, participants can still participate in the study on a volunteer basis.
* To be compensated for participation and be included in the main analysis, participants in study 3 must meet criteria for "struggling with distress" (ie, a score on either the depression or anxiety subscale greater than or equal to 3 (range 0-6), as these scores are suggestive of a depressive or anxiety disorder.

Exclusion Criteria:

* Having completed the study in the past
* Failing both of the attention checks in the baseline measures.
* Spending less than 3 minutes completing the study introduction and baseline measures (ie, were very likely bots)
* Indicating, at the end of the study, that one did not complete the study seriously and that one's data should not be included in analyses.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4370 (Actual)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Change in UCLA Loneliness Scale Version 3 at 8 weeks | Baseline, 8-week follow-up
  A 20-item measure of trait loneliness. Range 20-80 with higher scores indicated more severe loneliness. Included in studies 1, 3, and 4

SECONDARY OUTCOMES:
Change in UCLA Loneliness Scale Version 3 at 4 weeks | Baseline, 4-week follow-up
  A 20-item measure of trait loneliness. Range 20-80 with higher scores indicated more severe loneliness. Included in studies 1 and 3
Change in Depression Anxiety and Stress Scale - 9-item total score at 8 weeks | Baseline, 8-week follow-up
  A brief scale with subscales measuring depression, anxiety, and stress. Range 0-27 with higher scores indicating greater symptom severity. Included in all studies.
Change in Depression Anxiety and Stress Scale - 9-item total score at 4 weeks | Baseline, 4-week follow-up
  A brief scale with subscales measuring depression, anxiety, and stress. Range 0-27 with higher scores indicating greater symptom severity. Included in studies 1-3.
Change in 3-item Mini Social Phobia Inventory at 8 weeks | Baseline, 8-week follow-up
  A brief measure of social anxiety. Range 0-12 with higher scores indicating greater symptom severity. Included in studies 1 and 3
Change in 3-item Mini Social Phobia Inventory at 4 weeks | Baseline, 4-week follow-up
  A brief measure of social anxiety. Range 0-12 with higher scores indicating greater symptom severity. Included in studies 1 and 3
Change in Short form of the General Self-Efficacy Scale at 8 weeks | Baseline, 8-week follow-up
  A 6-item measure of general self-efficacy. Range 6-24 with higher scores indicating greater self-efficacy. Included in studies 1-3
Change in Short form of the General Self-Efficacy Scale at 4 weeks | Baseline, 4-week follow-up
  A 6-item measure of general self-efficacy. Range 6-24 with higher scores indicating greater self-efficacy. Included in studies 1-3
Change in Short form of the General Self-Efficacy Scale immediately post-intervention | Baseline, immediately post-intervention (roughly 30 minutes after beginning study for single-session conditions, and roughly 2 weeks after beginning study for 3-week iCBT condition)
  A 6-item measure of general self-efficacy. Range 6-24 with higher scores indicating greater self-efficacy. Included in studies 1-3.
Change in Beck Hopelessness Scale - 4-item at 8 weeks | Baseline, 8-week follow-up
  A brief version of a hopelessness measure. Range 4-12 with higher scores indicating more hopelessness. Included in all studies.
Change in Beck Hopelessness Scale - 4-item at 4 weeks | Baseline, 4-week follow-up
  A brief version of a hopelessness measure. Range 4-12 with higher scores indicating more hopelessness. Included in studies 1-3.
Change in Beck Hopelessness Scale - 4-item immediately post-intervention | Baseline, immediately post-intervention (roughly 30 minutes after beginning study for single-session conditions, and roughly 2 weeks after beginning study for 3-week iCBT condition)
  A brief version of a hopelessness measure. Range 4-12 with higher scores indicating greater hopelessness. Included in all studies.
Change in Frequency of actions and thoughts scale at 8 weeks | Baseline, 8-week follow-up
  A 12-item measure of adaptive thoughts and behaviors, improvement in which might be a target of cognitive behavioral therapy. Range 0-48 with higher scores indicating greater frequency of adaptive thoughts and behaviors. Included in all studies.
Change in Frequency of actions and thoughts scale at 4 weeks | Baseline, 4-week follow-up
  A 12-item measure of adaptive thoughts and behaviors, improvement in which might be a target of cognitive behavioral therapy. Range 0-48 with higher scores indicating greater frequency of adaptive thoughts and behaviors. Included in studies 1-3.
Program Feedback Scale | immediately post-intervention (roughly 30 minutes after beginning study for single-session conditions, and roughly 2 weeks after beginning study for 3-week iCBT condition)
  A 7-item measure of engagement with and acceptability of SSIs. Range 7-35 with higher scores indicating greater engagement with and acceptability of the SSI. Included in all studies.
Credibility and Expectancy Questionnaire | immediately post-intervention (roughly 30 minutes after beginning study for single-session conditions, and roughly 2 weeks after beginning study for 3-week iCBT condition)
  A 6-item measure of user-perceived intervention appeal and efficacy. Range 6-54 with higher scores indicating higher user-perceived intervention appeal and efficacy. Included in all studies.
Insight experience | immediately post-intervention (roughly 30 minutes after beginning study for single-session conditions, and roughly 2 weeks after beginning study for 3-week iCBT condition)
  A 1-item measure of whether one experienced an insight moment as a result of the program. Range 0-1 with 1 indicating presence of an insight experience and 0 indicating a lack of insight experience. Included in all studies.
Star rating | immediately post-intervention (roughly 30 minutes after beginning study for single-session conditions, and roughly 2 weeks after beginning study for 3-week iCBT condition)
  A rating of program quality, from 1-5 stars with more stars indicating greater quality. Included in all studies.
Change in PROMIS Meaning and Purpose in Life - 4-item at 4 weeks | Baseline, 4-week follow-up
  a 4-item measure of meaning and purpose in life. Range 4-20 with higher scores indicating a greater sense of meaning and purpose. Included in studies 2 and 3.
Change in PROMIS Meaning and Purpose in Life - 4-item at 8 weeks | Baseline, 8-week follow-up
  a 4-item measure of meaning and purpose in life. Range 4-20 with higher scores indicating a greater sense of meaning and purpose. Included in studies 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Schueller, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- Online (based at UC Irvine), Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared, including all measures. Participants' responses to open text response questions within the program will not be shared for the sake of privacy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available as soon as it is cleaned and de-identified and it will remain publicly available as long as possible.
Access Criteria: The data will be available to the public via an online dataset on the Open Science Framework (osf.io)

REFERENCES:
- [Background] Cacioppo JT, Cacioppo S. The growing problem of loneliness. Lancet. 2018 Feb 3;391(10119):426. doi: 10.1016/S0140-6736(18)30142-9. No abstract available. PMID 29407030
- [Background] Hickin N, Kall A, Shafran R, Sutcliffe S, Manzotti G, Langan D. The effectiveness of psychological interventions for loneliness: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Aug;88:102066. doi: 10.1016/j.cpr.2021.102066. Epub 2021 Jul 18. PMID 34339939
- [Background] Masi CM, Chen HY, Hawkley LC, Cacioppo JT. A meta-analysis of interventions to reduce loneliness. Pers Soc Psychol Rev. 2011 Aug;15(3):219-66. doi: 10.1177/1088868310377394. Epub 2010 Aug 17. PMID 20716644
- [Background] Kall A, Backlund U, Shafran R, Andersson G. Lonesome no more? A two-year follow-up of internet-administered cognitive behavioral therapy for loneliness. Internet Interv. 2020 Jan 17;19:100301. doi: 10.1016/j.invent.2019.100301. eCollection 2020 Mar. PMID 32071885
- [Background] Yamaguchi S, Ojio Y, Ando S, Bernick P, Ohta K, Watanabe KI, Thornicroft G, Shiozawa T, Koike S. Long-term effects of filmed social contact or internet-based self-study on mental health-related stigma: a 2-year follow-up of a randomised controlled trial. Soc Psychiatry Psychiatr Epidemiol. 2019 Jan;54(1):33-42. doi: 10.1007/s00127-018-1609-8. Epub 2018 Oct 12. PMID 30315333
- [Background] Rizvi SL, Finkelstein J, Wacha-Montes A, Yeager AL, Ruork AK, Yin Q, Kellerman J, Kim JS, Stern M, Oshin LA, Kleiman EM. Randomized clinical trial of a brief, scalable intervention for mental health sequelae in college students during the COVID-19 pandemic. Behav Res Ther. 2022 Feb;149:104015. doi: 10.1016/j.brat.2021.104015. Epub 2021 Dec 21. PMID 34958980
- [Background] Murphy ST, Frank LB, Chatterjee JS, Baezconde-Garbanati L. Narrative versus Non-narrative: The Role of Identification, Transportation and Emotion in Reducing Health Disparities. J Commun. 2013 Feb;63(1):10.1111/jcom.12007. doi: 10.1111/jcom.12007. PMID 24347679
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Derived] Kaveladze BT, Gastelum SF, Ngo DC, Delacruz P, Cohen KA, Kall A, Andersson G, Schleider JL, Schueller SM. A randomized controlled trial comparing brief online self-guided interventions for loneliness. J Consult Clin Psychol. 2025 Jan;93(1):54-63. doi: 10.1037/ccp0000908. Epub 2024 Sep 26. PMID 39325409

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT05687162/Prot_SAP_001.pdf